CLINICAL TRIAL: NCT06947239
Title: Additional Effects of Mirror Therapy on Shoulder Mobility and Function in Post-stroke Adhesive Capsulitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/67
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Range of Motion; Adhesive Capsulitis; Mirror Therapy
Keywords: post stroke patients; Range of motion correction; mirror therapy exercises
MeSH Terms: conditions — Bursitis | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror therapy along with conventional therapy (Experimental): It includes participants receiving mirror therapy session in adhesive capsulitis of post stroke patients for a period of 6 weeks.
  The experimental group will receive 20 minutes of conventional therapy followed by 20 minutes of mirror therapy training including 3 minutes of rest period between the interventions.
  Interventions: Procedure: Mirror therapy along with conventional therapy
- Conventional Therapy (Active Comparator): it includes 11 participants receiving conventional physical therapy for a period of 6 weeks. The control group will receive the conventional therapy for 40 minutes including:
  1. Heat pack & TENS to alleviate pain for 15 minutes
  2. Shoulder isometric exercises 10 reps
  Interventions: Procedure: Control Group

INTERVENTIONS:
Procedure: Mirror therapy along with conventional therapy — The experimental group will receive 20 minutes of conventional therapy followed by 20 minutes of mirror therapy training including 3 minutes of rest period between the interventions.
  WEEK OF INTERVENTION:
  TASK PERFORM IN FRONT OF MIRROR:
  WEEK :1-2
  ACTIVE SHOULDER ROM:
  flexion, abduction, external-internal rotation movements of the intact extremity
  Increase the number of repetition according to the patient progression
  WEEK:3-4
  ACTIVITIES TARGETING SHOULDER ROM:
  Cleaning the mirror with a towel(internal rotation+ abduction)
  Lifting a glass to drink ( flexion + abduction)
  Holding a brush to comb hair (external rotation
  WEEK:5-6
  Overhead reaching
  (pasting stickers on the
  mirror)(internal rotation
  / abduction)
  Lifting a bottle overhead.
  ( flexion/abduction)
  Throwing a ball (external
  rotation)
  PROGRESSION OF TASK SPECIFIC MIRROR THERAPY:
  WEEK: 1-2 Increase the number of repetition according to the patient progression WEEK:3-4 Add water in glass Transfer glass
  Arms: Mirror therapy along with conventional therapy
Procedure: Control Group — Details: Weeks wise:
  The control group will receive 20 mints of conventional therapy .
  1. Heat pack & TENS to alleviate pain for 15 minutes
  2. Shoulder isometric exercises 10 reps
  3. Active and passive Range of Motion exercises 10 reps each
  4. Codman exercises 10 reps each
  5. Wand exercises 10 reps each
  Arms: Conventional Therapy

SUMMARY:
The estimated annual incidence of stroke in Pakistan is 250/100, 000. Upper limb impairments and post-stroke musculoskeletal complications such as pain, subluxation and restricted joint range of motion are commonly reported. Among many other shoulder impairments, adhesive capsulitis is a leading cause of limited mobility, reduced range of motion, and pain in stroke patients.

The aim of the current study will benefit the clinicians and physiotherapists as it provide an insight to treat post stroke adhesive capsulitis. Effects of mirror therapy have been established but the literature does not provide best treatment approaches or modalities for different types of Hemiplegic shoulder pain. This study will address the limitations in treatment approaches concerning the shoulder joint and its mobility in post-stroke adhesive capsulitis.

The study will be non-blinded randomized control trial, consisting of two groups. Study will be conducted over a period of 1 year. Subjects will be selected via non-probability purposive sampling technique using coin toss method followed by randomization into two groups (A and B).Ethical approval will be obtained from ERC FUMC.

One group will receive mirror therapy while other will receive conventional exercises treatment for period of 6 weeks. Baseline tests will be performed before and after the intervention of mirror therapy & outcome measure assessments will be done after every 3 weeks for a total period of 6 weeks intervention period. Data will be entered and analyzed on SPSS version 22.

DETAILED DESCRIPTION:
OBJECTIVES OF STUDY

1. To determine the effects of mirror therapy along with conventional therapy on improving shoulder joint range of motion in post-stroke adhesive capsulitis patients.
2. To determine the effects of mirror therapy along with conventional therapy on improving shoulder joint function in post-stroke adhesive capsulitis patients.
3. To compare the difference between the effects of mirror therapy with conventional therapy alone for improving shoulder mobility and function in post stroke adhesive capsulitis patients.

HYPOTHESIS ALTERNATE HYPOTHESIS

1. There is a statistically significant effect of mirror therapy in improving the shoulder joint Range Of Motion in post-stroke adhesive capsulitis patients. (p > 0.05).
2. There is a statistically significant effect of mirror therapy in improving the shoulder joint function in post-stroke adhesive capsulitis patients. (p > 0.05).

NULL HYPOTHESIS

1. There is a statistically significant effect of mirror therapy in improving the shoulder joint Range Of Motion in post-stroke adhesive capsulitis patients. (p > 0.05).
2. There is a statistically significant effect of mirror therapy in improving the shoulder joint function in post-stroke adhesive capsulitis patients. (p > 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Both genders male and female
* Age 40-70 years
* Ability to understand and follow simple verbal instructions
* Patients able to stand for at least 10-15 mins.
* Ability to participate in a therapy session by coming to hospital.
* Chronic Stroke (ischemic) patients (6 months-1year) with adhesive capsulitis (capsular pattern :external rotation> abduction > internal rotation)
* Scores of >24 on Montreal Cognitive assessment scale.

Exclusion Criteria:

* Upper limb fractures or cervical spine pathology or radiculopathy
* History of upper limb surgery or trauma
* Rotator cuff pathology or prolonged immobilization of upper limb
* Rheumatic disease, fibromyalgia or any other musculoskeletal disorder that is altering upper extremity movement
* Any other neurological condition

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Range of motion | 6 weeks
  Goniometer will be used to assess range of motion at the shoulder
cognitive impairment | 6 weeks
  Montreal cognitive assessment test that was used to detect mild cognitive impairment

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan